CLINICAL TRIAL: NCT02927574
Title: Drug Or No Drug (DOND): Systematic Review and Meta-Analysis on Drug-Coated Balloon Angioplasty (DCB) vs. Plain Old Balloon Angioplasty (POBA) in De-novo Femoropopliteal Disease
Brief Title: Systematic Review and Meta-Analysis on DCB vs. POBA in De-novo Femoropopliteal Disease
Acronym: DOND
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Ulf Teichgräber, Prof. Dr. med., Jena University Hospital
Other Study IDs: IDIR/005/2016
Record Dates: First submitted 2016-09-01; First posted 2016-10-07 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: drug-coated balloon angioplasty; angioplasty; plain old balloon angioplasty; peripheral arterial disease; intermittent claudication; systematic review; meta-analysis; Paclitaxel
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DCB: Treatment with Paclitaxel drug-coated balloon angioplasty (DCB)
  Interventions: Device: DCB
- POBA: Treatment with plain old balloon angioplasty (POBA)
  Interventions: Device: POBA

INTERVENTIONS:
Device: DCB
  Groups: DCB
Device: POBA
  Groups: POBA

SUMMARY:
Restenosis is still an issue after endovascular revascularization for femoropopliteal occlusive disease. One approach to reduce the rates of restenosis and reintervention is local application of Paclitaxel with drug-coated balloon angioplasty. The purpose is to conduct a systematic review and meta-analysis of randomized-controlled trials comparing on Drug-Coated Balloon angioplasty (DCB) vs. Plain Old Balloon Angioplasty (POBA) in de-novo femoropopliteal disease.

DETAILED DESCRIPTION:
Peripheral arterial disease is the third leading entity of atherosclerosis. The femoropopliteal segment is affected in most patients. Endovascular revascularisation is one possible treatment option, but high rates of restenosis, especially in complex lesions, are a limiting factor. Bare-metal stents failed to show a long-term superiority in a Cochrane systematic review. Another approach to prevent restenosis is local delivery of an antiproliferative drug (e.g. Paclitaxel) via Drug-Coated Balloon Angioplasty. New studies did report their results since the publication of earlier meta-analyses. It's time for an up-to-date systematic review. Prior systematic reviews did not address risk of bias nor did they take differences in treatment strategy despite the used balloon catheter into consideration.Some previous reviews did compare results from different points in time, e.g. analysis of 6 months' results together with 24 months' results.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials
* DCB vs. POBA
* focus on de-novo femoropopliteal lesions
* registration in a clinical trials registry
* available study protocol (either in clinical trial registry or published)

Exclusion Criteria:

* non-randomized controlled trials
* focus on below-the-knee interventions
* focus on iliac artery interventions
* focus on treatment of critical limb ischemia
* focus on treatment of in-stent restenosis
* usage of additional devices except for bare-metal stent (e.g. atherectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with intermittent claudication due to de novo femoropopliteal peripheral arterial disease.
Sampling Method: Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Freedom from (clinical driven) Target Lesion Revascularisation (FfTLR) | 12 months
  Freedom from repeated intervention of the index lesion (due to binary restenosis > 50% and/or recurrent symptoms)
Freedom from (clinical driven) Target Lesion Revascularisation (FfTLR) | 24 months
  Freedom from repeated intervention of the index lesion (due to binary restenosis > 50% and/or recurrent symptoms)

SECONDARY OUTCOMES:
Primary Patency (PP) | 12 and 24 months
  freedom from repeated intervention (FfTLR) and freedom from binary restenosis > 50% [comment: The metaanalysis compares the endpoints of different trials comparing DCB vs. POBA. The primary patency is a commonly used efficacy endpoint in those trials; information on this endpoint will be extracted from already published trial data.]
Secondary Patency (SP) | 12 and 24 months
  freedom from binary restenosis after
  1. single repeated endovascular revascularization or
  2. no repeated Intervention [comment: The metaanalysis compares the endpoints of different trials comparing DCB vs. POBA. The secondary patency is another commonly used efficacy endpoint in those trials; information on this endpoint will be extracted from already published trial data.]
Late Lumen Loss (LLL) | 6 and 12 months
  Difference of minimal lumen diameter at follow-up compared to minimal lumen diameter after index procedure
ABI | 12 and 24 months
  Ankle-Brachial-Index
Rutherford-Becker Classification | 12 and 24 months
  Clinical stage of disease according to Rutherford-Becker Classification
Functional outcome | 12 and 24 months
  Functional result eg. Walking Impairment Questionnaire (WIQ) or treadmill test
Quality of Life (QoL) | 12 and 24 months
  Quality of Life outcome eg. EQ5D

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Teichgräber, Prof., Principal Investigator — University Hospital Jena